CLINICAL TRIAL: NCT07216885
Title: Solv Multi-Pass Hemodialysis System In-Center Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT22047
Record Dates: First submitted 2025-10-06; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Solv Multi-Pass Hemodialysis System In-Center Subjects (Experimental): All subjects enrolled in the study and treated with the Solv Multi-Pass Hemodialysis System
  Interventions: Device: Solv Multi-Pass Hemodialysis System

INTERVENTIONS:
Device: Solv Multi-Pass Hemodialysis System — Solv Multi-Pass Hemodialysis System

SUMMARY:
Solv In-Center clinical study is a pre-market, prospective, multicenter, single arm, open-label clinical study. The patient population will include patients with kidney failure or insufficiency requiring hemodialysis and/or ultrafiltration. Eligibility will be open to incident dialysis patients and patients currently receiving HD in an in-center environment. All vascular access types including AV-fistula, AV-graft, and tunneled hemodialysis catheters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able and willing to give Informed Consent and interested to participate in the study
* Subject aged 18 years or older
* Subjects meets one of the following three conditions:

  * End stage renal disease (ESRD) patients who have been adequately treated with maintenance HD and deemed stable, according to the investigator, for at least three months
  * Incident end stage renal disease (ESRD) patients who have been prescribed HD therapy
  * Subjects on peritoneal dialysis who require conversion to hemodialysis, according to the investigator
* Subjects who have adequate access, capable of providing a blood flow rate of at least 300 mL/min
* Subject understands the nature of the procedures and the requirements of the study protocol
* Subject is willing and able to comply with the protocol requirements and return to the treatment center for all required treatments and clinical evaluations

Exclusion Criteria:

* Subjects with baseline dry weight of ≤ 60 kg or ≥ 110 kg
* Subjects with a documented history of non-compliance to scheduled hemodialysis sessions or clinic visits
* Subjects who are pre-scheduled for a living kidney transplant within the next two months, who plan a change to peritoneal dialysis (PD) within the next two months or who require single needle dialysis therapy
* Subjects with unstable electrolytes or acid base balance, in the opinion of the investigator
* Subjects with any major surgery or major adverse cardiac event within 3 months of screening
* Subjects with hemodynamic instability, defined as repeated hypo/hypertension, in the past 30 days from screening
* Subjects with active or ongoing infection, in the opinion of the Investigator
* Subjects with known Hepatitis B, C or HIV infection
* Subject with documented coagulation disorders, active or bleeding risk or who is intolerant to heparin
* Subjects who are currently participating or have previously participated in another interventional clinical trial in the past 4 weeks from screening
* Subjects with any comorbidities possibly conflicting with the study purpose or procedures, in the opinion of the Investigator
* Subjects who are pregnant or lactating or any patient with a childbearing potential who refuses to use medically acceptable means of contraception
* Subjects with an active, malignant disease and whose life expectancy is < 6 months, in the opinion of the investigator
* Subjects with a hemoglobin < 9 gm/dl in the past 30 days from screening
* Subjects with significant intradialytic hypotension in 30 days from screening
* Subjects with shock within 30 days from screening
* Subjects with active seizures in the last 6 months from screening
* Subjects with history of hemolytic anemia or thrombocytopenia
* Subjects with vascular access dysfunction (switching ports (reverse lines or catheter replacement) in 30 days prior to screening, multiple tPA (tissue plasminogen activator) administrations) or patient who has had a thrombectomy procedure within 30 days prior to screening
* Subjects with a documented history of congestive heart failure with symptoms consistent with NYHA Class III or IV, according to the investigator, or documented severe left ventricular dysfunction
* Subjects with fluid overload due to intractable ascites secondary to liver cirrhosis
* Subjects with active, life-threatening rheumatologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | through study completion, an average of 1 year
  Evaluate the number of serious device-related adverse events that occur during the In-Center Phase of the study, to confirm there are no additional risks associated with the Solv System implementation of sorbent-based HD.
  Events listed below contribute to the primary safety endpoint and include all serious device-related adverse events.
Primary Performance Endpoint | through study completion, an average of 1 year
  Evaluate the mean single pool (sp)Kt/V for subjects undergoing conventional In-Center HD with the Solv Multi-Pass Hemodialysis System during the eight-week study Phase.

SECONDARY OUTCOMES:
Serious adverse events and all device and/or therapy related adverse events | through study completion, an average of 1 year
  Quantify all serious adverse events and all device and/or therapy related adverse events which occur during the Run-in and In-Center Phase, regardless of relationship to the Solv Multi-Pass Hemodialysis System or seriousness
Uremic toxin profile | through study completion, an average of 1 year
  Characterize uremic toxin profile of urea, β-2 microglobulin and myoglobin
Electrolyte balance and evaluate mineral metabolism | through study completion, an average of 1 year
  Verify electrolyte balance and evaluate mineral metabolism by characterizing pre-post session sodium, chloride, potassium, calcium, magnesium, bicarbonate, phosphate and glucose
Nutritional status | through study completion, an average of 1 year
  Evaluate nutritional status by characterizing pre-post session albumin and change in body mass index (BMI)
Inflammation markers | through study completion, an average of 1 year
  Assess inflammation markers by characterizing pre-session values of C-reactive protein (CRP)
Volume of UF removed | through study completion, an average of 1 year
  Confirm that the volume of UF removed as indicated by the Solv System will be within 10% of target UF volume entered into the device per session, accounting for prescribed estimated dry weight, treatment time, and rinse back volume
Use of intradialytic medications | through study completion, an average of 1 year
  Summarize the use of intradialytic anticoagulants and erythropoietin, phosphate binders and iron doses
Patient-reported outcome measures with KDQOL-36 | through study completion, an average of 1 year
  Quantify patient-reported outcome measures on KDQOL-36 questionnaire to assess patient quality of life and satisfaction, along with physicial and mental health. The KDQOL will be collected at baseline and IC- weeks 1, 4, and 8 for comparison
Patient-reported outcome measures with Dialysis Recovery Time Questionnaire | through study completion, an average of 1 year
  Quantify patient-reported outcome measures on dialysis recovery time to assess amoujnt of time it takes for each subject to recover from a dialysis session. The DRT questionnaire will be collected at baseline and In-Center Weeks 1, 4, & 8 for comparison.
User Experience with Solv | through study completion, an average of 1 year
  Characterize the user experience via questionnaire (e.g., Solv set-up, recharging process, alarm management). The questionnaire will be provided to a sampling of users.